CLINICAL TRIAL: NCT06909448
Title: Effect of Capacitive and Resistive Radiofrequency on Postpartum Diastasis Recti
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Gamil Omar, assistant lecturer, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: radiofrequency on diastasis
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Diastasis Recti Abdominis (DRA); Radiofrequency
Keywords: Diastasis recti, radiofrequency therapy, physical exercises, postpartum
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator): It will be consisted of 40 postpartum women who will only wear abdominal belt for 14 weeks.
  Interventions: Device: abdominal belt
- study group (Active Comparator): will wear the same abdominal belt for 6 weeks then participating in TECAR therapy 3 sessions /week for 8 weeks.
  Interventions: Device: abdominal belt; Device: TECAR therapy

INTERVENTIONS:
Device: abdominal belt — 40 postpartum women will only wear abdominal belt for 14 weeks.
Device: TECAR therapy — will wear the same abdominal belt for 6 weeks then participating in TECAR therapy 3 sessions /week for 8 weeks.
  Arms: study group

SUMMARY:
To evaluate the effect of capacitive and resistive radiofrequency on postpartum rectus abdominis diastasis.

DETAILED DESCRIPTION:
Eighty females postpartum with rectus diastasis will be included in this study; they will be recruited the outpatient clinic at El Mahalla Al Kobra (The first author's pervious workplace) and will be referred by obstetric and genecology physicians. Patients will be assigned into two groups.

Group A: It will include 40 patients participating in abdominal belt. Group B: It will include 40 patients participating in abdominal belt plus TECAR therapy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Postpartum women (7 days after delivery) having diastasis recti (separation between the two recti more than 2.5cm at the level of umbilicus).

  2. Multiparous women (2-3) times delivered vaginally with or without episiotomy.

  3. Their age will be ranged from 20 -35 years old. 4. Their BMI will be less than 30 kg/cm2.

Exclusion Criteria:

* Any participant will be excluded if she meets one or more of the following criteria:

Postpartum women will be excluded from the study if they have:

1. Abdominal or back surgery.
2. Abdominal hernia.
3. History of abnormal pregnancy, uterine fibroid or polyhydramnios during pregnancy.
4. Neurological disorders as multiple sclerosis, stroke and spinal lesion.
5. Musculoskeletal diseases such as fractures muscle strains, severe knee osteoarthritis which may affect their physical activity.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-04-06 (Estimated); Primary Completion 2025-07-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Ultrasound | 14 week
  The distance between the recti muscles at 3 levels will be measured at the beginning and again at the end of the study duration, i.e., 8 weeks. The desired measurement locations will be marked with a water-soluble pen: 4.5 cm above the umbilicus, at the midpoint, and 4.5 cm below the umbilicus. The measurements will be performed at rest and during contraction. Each woman will be asked to lie in a crock lying position, crossing the arms over the chest and raising the head until the spine of the scapulae will be off the table surface. The women will maintain a partial curl-up while the examiner palpates the medial borders of the right and left rectus abdominis muscle bellies at the marked location. With the linear transducer, it will be positioned transversely along the linea alba in the direction of the muscles and adjusted to perceived inert recti distance width. Three trials will be taken for each assessment, and the mean will be recorded. (Khandale & Hande, 2016).
trunk flexors strength and endurance | 14 week
  Trunk flexion strength will be graded from zero to five using Daniels and Worthingham's procedure (Hislop et al., 2013) as follows:
  Grades: (Hislop et al., 2013). Grade 5 (Normal) Patient complete ROM until inferior angle of the scapulae are off table (weight of arms serves as resistance).
  Grade 4 (Good) Patient complete ROM until inferior angle of the scapulae are off table. Resistance of arms is reduced in the cross-chest position.
  Grade 3 (Fair) Patient complete ROM and lifts trunk until inferior angle of the scapulae are off table with arms at side.
  Grade 2 (Poor) Patient is unable to clear the inferior angle of the scapula from the table Grade 1 (Trace) No depression of the rib cage but visible or palpable contraction occurs.
  Grade 0 (Zero) No activity
  Patient Positioning:
  Grade 5 (Normal): Supine with fingertips lightly touching the back of the head. For grade 4: Supine with arms crossed over chest. For grade 3: Supine with arms at side. For grade 0 to 2: Supine with arms at
Assessment of functional status | 14 week
  All participating women with diastasis recti in both groups (A&B) will be asked to fill the Inventory of functional status after childbirth questionnaire before and after the end of the study program.

IPD SHARING:
Plan to Share IPD: No